CLINICAL TRIAL: NCT01430312
Title: A Randomized, Double-blind, Vehicle-controlled Phase 1 Dermal Safety Study Using a 21 Day Cumulative Irritant Patch Test Design to Evaluate the Local Tolerability of Azelaic Acid Pre-Foam Formulation in Healthy Volunteers
Brief Title: 21 Day Irritancy Test of Azelaic Acid Pre-foam Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15853; 1401841 (Other: Company internal)
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2014-02

CONDITIONS: Healthy
Keywords: dermal irritative potential
MeSH Terms: interventions — Water; Sodium Dodecyl Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Verum (Experimental): Topical application of verum (azelaic acid pre-foam formulation) on the skin
  Interventions: Drug: azelaic acid pre-foam formulation
- Vehicle (Placebo Comparator): Topical application of vehicle formulation (same as verum but without active drug substance) on the skin
  Interventions: Drug: Vehicle pre-foam formulation
- Negative control (Placebo Comparator): Topical application of distilled water (negative control) on the skin
  Interventions: Drug: Water
- Positive control (Active Comparator): Topical application of 0.5% Sodium Lauryl sulfate (positive control) on the skin
  Interventions: Drug: Sodium lauryl sulfate

INTERVENTIONS:
Drug: azelaic acid pre-foam formulation
  Arms: Verum
Drug: Vehicle pre-foam formulation
  Arms: Vehicle
Drug: Water
  Arms: Negative control
Drug: Sodium lauryl sulfate
  Arms: Positive control

SUMMARY:
The purpose of this study is to determine the irritancy potential of azelaic acid pre-foam formulation.

DETAILED DESCRIPTION:
This is the standard patch test over 21 days of exposure of the test product,its vehicle and a positive as well as a negative control.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* male ore female subjects
* aged 18 - 65 years
* ability to understand and fulfill the study requirements

Exclusion Criteria:

* affected skin in designated test area
* pregnancy or lactation
* not willing to comply with study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
irritancy rating scale | 21 days
  skin reaction as well as superficial layer effects will be scored according to standardized scales

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Robert I. Cooper, MD, Fargo, North Dakota, United States